CLINICAL TRIAL: NCT07339189
Title: Piloting AI-Delivered Dialectical Behavioral Therapy for Suicide Prevention in Older Patients Living With HIV
Brief Title: HIV Suicide Prevention With AI-DBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Elissa Kozlov, Ph.D, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO2024000600; R34MH134693 (NIH)
Record Dates: First submitted 2026-01-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Ideation and Behavior; HIV; AIDS (Acquired Immune Deficiency Syndrome)
Keywords: suicide; HIV; mHealth
MeSH Terms: conditions — Suicidal Ideation; Behavior; Acquired Immunodeficiency Syndrome; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care (No Intervention): Usual care
- AI-DBT (Experimental): AI-DBT group will receive 14 videos under 5 minutes across 7 weeks and the opportunity to engage in skills coaching with an AI chatbot
  Interventions: Behavioral: AI-DBT

INTERVENTIONS:
Behavioral: AI-DBT — Participants will receive 14, 5 minute videos delivered 2x/week that describe DBT skills and tools. They will also receive the option of engaging in coaching sessions.
  Arms: AI-DBT

SUMMARY:
One in four older persons living with HIV/AIDS (PLWHA) report at least one suicide attempt in their lifetime, and the risk for death by suicide is 100 times higher in PLWHA than in the general population. Currently, there are no behavioral interventions that specifically address suicide prevention for older PLWHA, despite their unique biopsychosocial and structural risk factors. Through this work, investigators will adapt Dialectical Behavior Therapy, an evidence-based intervention for suicide prevention, for patients with PLWHA to be delivered by an AI-powered conversational Agent developed by our industry partner, Empower Health. Investigators will then pilot test the feasibility, usability, acceptability and preliminary efficacy to improve self-efficacy to manage negative emotions in n=50 older adults living with HIV/AIDS.

DETAILED DESCRIPTION:
One in four older persons living with HIV/AIDS (PLWHA) report at least one suicide attempt in their lifetime, and the risk of death by suicide is 100 times higher in PLWHA than in the general population. In the United States, there are approximately 1.2 million PLWHA, and 35% are adults aged 55 and over. Older PLWHA experience unique combinations of stressors including externalized and internalized stigma from advanced age and disease status. Despite the increased risk and unique risk factors older PLWHA have for suicide mortality, there have been no interventions developed specifically for this population to address suicide risk. Dialectical Behavioral Therapy (DBT) shows significant impact at reducing suicidal behaviors by improving one's self-efficacy to manage negative emotions. DBT has never been evaluated with PLWHA for suicide prevention, representing a critical gap in the science. Innovative solutions to mental health care, such as AI-powered chatbots, have also not been studied extensively in older PLWHA. The objective of this R34 Intervention Development and Pilot grant proposal is to adapt DBT Skills and Coaching for suicide prevention in older PLWHA to be delivered via brief videos and Angel. Angel is an artificial intelligence (AI)-powered conversational agent developed by CareAngel, a company that leverages cutting edge AI and natural language processing technology. Investigators plan to adapt existing evidence-based DBT skills videos and add coaching support from Angel in a 6-week intervention with older PLWHA. This proposal has the following specific aims: Phase 1: Adaptation: Aim 1) To adapt DBT Skills and Coaching for PLWHA seeking care in infectious disease practices to be delivered via Angel. Phase 2: Pilot feasibility and preliminary efficacy RCT with n=50 PLWHA: Aim 2) To establish the feasibility, acceptability, and usability of the adapted DBT Skills and Coaching intervention through key metrics of use, survey item responses, and qualitative interviews surrounding barriers and facilitators to use with patients enrolled in the intervention. Aim 3) To explore the preliminary efficacy, relative to usual care control, of DBT skills videos and Angel-delivered DBT Coaching on the target mechanism, self-efficacy to manage negative emotions, as well as exploratory clinical outcomes including suicide outcomes, mood, and medical treatment adherence. This proposed work is of high scientific and public health significance for numerous reasons: 1.) older PLWHA have elevated suicide risk. 2.) there is a paucity of suicide prevention intervention research for PLWHA. 3.) while Dialectical Behavioral Therapy has been studied in over 30 randomized controlled trials with demonstrated efficacy to improve psychological outcomes in diverse populations, to our knowledge, this intervention has never been piloted with older PLWHA. 4.) Innovative solutions to mental health care, such as AI-powered chatbots + videos, have not been studied in older PLWHA, thus this proposal represents an exciting opportunity to fill critical gaps in the literature on potentially scalable, implementable, and effective approaches to suicide prevention in PLWHA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50+
* evidence of suicide risk as defined by at least one of the following: PHQ-9 suicide item > 0, Ask Suicide Questions (ASQ, an NIMH-supported suicide risk screener with a version tailored for primary care) > 0, expression of suicidal thoughts to the provider during appointment, a suicide attempt in the past year, or PHQ-9 total score ≥ 8,
* ability to read and communicate fluently in English or Spanish
* not at imminent risk for suicide (does not have significant intent to die within 48 hours)
* has a smartphone capable of texting and accessing the internet.

Exclusion Criteria:

* deemed clinically inappropriate to participate because of severe psychosis, severe substance use, or severe cognitive deficits that would interfere with their comprehending study and intervention material.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy to manage emotions | baseline, 6 and 12 weeks for long-form.
  Scale to determine if someone has self-efficacy to manage negative emotions

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Kozlov, PhD, Principal Investigator — Rutgers
Locations (2):
- United States (2):
  - New Jersey Community Research Initiative, Newark, New Jersey
  - RWJB Infectious Disease, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No
The plan is to share data with the NIMH NDA repository.